CLINICAL TRIAL: NCT02198001
Title: Prospective Randomized Clinical Study: Role of Platelet Rich Fibrin (PRF) in the Tooth Extraction Site in the Prevention of Jaw Osteonecrosis on Patients Under Bisphosphonates Therapy
Brief Title: Prospective Randomized Study: Assessment of PRF Efficacy in Prevention of Jaw Osteonecrosis After Tooth Extraction
Acronym: PRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B403201318408
Record Dates: First submitted 2014-07-15; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Bisphosphonate-Associated Osteonecrosis of the Jaw
Keywords: Platelets; fibrin; growth factors; bisphosphonates; tooth extraction
MeSH Terms: conditions — Bisphosphonate-Associated Osteonecrosis of the Jaw | interventions — Tooth Extraction; Anti-Bacterial Agents; Amoxicillin-Potassium Clavulanate Combination; Clindamycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tooth extraction and insertion of PRF (Active Comparator): Experimental: Atraumatic tooth extraction with antibiotics( amoxicillin clavulanate combination) .Insertion of PRF membrane in tooth-extraction site.
  Interventions: Drug: tooth extraction with antibiotics (amoxicillin- clavulanate, clindamycine); Procedure: atraumatic extraction
- No PRF (Placebo Comparator): Atraumatic extraction with antibiotic without PRF insertion
  Interventions: Drug: tooth extraction with antibiotics (amoxicillin- clavulanate, clindamycine); Procedure: atraumatic extraction

INTERVENTIONS:
Drug: tooth extraction with antibiotics (amoxicillin- clavulanate, clindamycine) — BPs per os< 3ans: amoxicillin- clavulanate J-1 à J+10
  BPs IV ou per os> 3ans ou per os + comordibities (diabetes, immunosuppression, tobacco):
  amoxicillin- clavulanate J-3 à J+10
  In case of allergy:
  BPs per os: clindamycine J-1 à J+10
  BPs IV ou per os> 3ans ou per os + comordibities (diabetes, immunosuppression, tobacco):
  clindamycine J-3 à J+10
  Other Names: antibiotherapy before and after extraction
Procedure: atraumatic extraction — Atraumatic tooth extraction, alveolar bone reduction, hermetic mucosal closure
  Other Names: - atraumatic tooth extraction; - hermetic mucosal closure

SUMMARY:
This prospective study will include patients taking or having taken bisphosphonates and needing dental extractions.

The aim of this study is to validate the contribution of PRF (Platelet Rich Fibrin) in tooth extraction sites.

In the test group (PRF) and in the control group (no PRF), we use the same atraumatic extraction protocol associated with the same antibiotic procedure.

DETAILED DESCRIPTION:
Dental extractions are the main cause of jaw osteonecrosis in patients taking oral or iv bisphosphonates.

This prospective randomized study will include a cohort of 100 patients treated with bisphosphonates (for benign or malignant conditions) and requiring dental extractions (non-retainable teeth for infectious, traumatic or parodontal reasons). 50 patients will benefit of PRF placement in the tooth extraction site (group 1) while 50 patients do not (group 2).

The rest of the procedure will be the same in the 2 arms. In the literature, studies suggest a benefit from a long term antibiotherapy before and after tooth extraction. Extraction procedure should be the least traumatic as possible.

The main objective of our study is to assess, after tooth extraction, the contribution of PRF in the prevention of jaw osteonecrosis induced by bisphosphonates.

A follow-up period of one year after extraction is indicated.

ELIGIBILITY:
Inclusion Criteria:

* patients taking bisphosphonates whatever the indication, the type, the administration and the duration of treatment (we include patients taking or having taken bisphosphonates, even several years ago)
* And who need tooth extraction (not recoverable in conservative dentistry and symptomatic tooth: dental and periodontal infections, symptomatic traumatic tooth fracture).

Exclusion Criteria:

* pregnant women
* younger than 50 years old
* jaw's radiotherapy
* history of jaw osteonecrosis
* jaw metastasis from an other cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Number of jaw osteonecrosis after tooth extraction | 1year
  7 symptoms > 6 weeks for the diagnosis of osteonecrosis:
  * bone exposure
  * bone spicule
  * mucosal inflammation
  * pain
  * paresthésias
  * suppuration
  * jaw fracture
    * number of jaw osteonecrosis after tooth extraction in the oral bisphosphonates group in comparison with the IV bisphosphonates group

OTHER OUTCOMES:
Contribution of comorbidities factors in the appearance of osteonecrosis | 1 year
  comorbidities:
  * diabetes,
  * immunosuppression (corticoids, chemotherapy, immunosuppressive treatment)
  * tobacco
Number of days in tooth-extraction healing in the two groups | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Hervé P Reychler, MD, DMD, Study Chair — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (3):
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - Centre Hospitaliser Ambroise Paré, Mons
  - Clinique et maternité Sainte Elisabeth, Namur

REFERENCES:
- [Derived] Beth-Tasdogan NH, Mayer B, Hussein H, Zolk O, Peter JU. Interventions for managing medication-related osteonecrosis of the jaw. Cochrane Database Syst Rev. 2022 Jul 12;7(7):CD012432. doi: 10.1002/14651858.CD012432.pub3. PMID 35866376